CLINICAL TRIAL: NCT05237557
Title: Impact of an Operating Room Nurse Pre-operative Dialogue on Anxiety, Satisfaction and Early Postoperative Outcomes in Patients Undergoing Major Visceral Surgery - a Single Center, Open-label, Randomized Controlled Trial
Brief Title: Impact of an Operating Room Nurse Pre-operative Dialogue in Patients Undergoing Major Visceral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolas DEMARTINES (Other)
Responsible Party: Sponsor-Investigator, Nicolas DEMARTINES, Head of Visceral Surgery Department, Professor of Surgery, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-00202
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Anxiety; Post Operative Pain; Postoperative Nausea; Postoperative Complications; Satisfaction, Patient
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Complications; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Single center, Open-label, Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental)
  Interventions: Behavioral: Preoperative nurse dialogue
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Preoperative nurse dialogue — Performance of a preoperative nurse dialogue prior major visceral surgery
  Arms: Interventional group

SUMMARY:
Single-center, open label, randomized controlled trial of a preoperative nursing dialogue in patient undergoing major visceral surgery aiming in evaluating its impact on patients' anxiety, satisfaction and early postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective major visceral surgery
* Hospitalization the day before surgery
* Sufficient command of French language

Exclusion Criteria:

* emergency procedures (after unplanned admission)
* inability to obtain informed consent or refusal
* inability to follow intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | 5-10 minutes after intervention
  State-Trait Anxiety Inventory Form Y (STAI-Y)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Visceral Surgery, University Hospital CHUV, Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No